CLINICAL TRIAL: NCT02094326
Title: A Retrospective, Multicentre Observational Study to Assess the Management of Synthetic Disease-modifying Antirheumatic Drug (DMARD) at the Onset of Adverse Events, Intolerance or Lack of Efficacy in Real Life in Patients With Rheumatoid Arthritis
Brief Title: Study to Assess the Management of Synthetic Disease-modifying Antirheumatic Drug (DMARD) at the Onset of Adverse Events, Intolerance or Lack of Efficacy in Rheumatoid Arthritis (RA)
Acronym: SAR-FAME
Status: Completed | Type: Observational
Sponsor: Fundación Andaluza de Reumatología (Other)
Responsible Party: Sponsor
Other Study IDs: SAR-FAM-2013-01
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find patterns in the use of non-biological DMARDs as the initial treatment of RA and how adverse events (AEs), intolerance or lack of efficacy may impact therapeutic decisions in real life in the Spanish Andalusian region.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes ≥ 18 years.
* Patients diagnosed with RA (according to the American College of Rheumatology (ACR) 2010 criteria) between January 2008 and December 2012 and who have initiated treatment with at least one synthetic DMARD during that period.
* Patients who have given written informed consent for their data to be collected and reviewed.

Exclusion Criteria:

* Patients who are already participating in a clinical trial/s at the moment of participation in this study.
* Patients with whom it is suspected there will be insufficient information to complete the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Navarro, Dr., Study Director — Fundacion Andaluza de Reumatologia
Locations (11):
- Spain (11):
  - Hospital Reina Sofía, Córdoba, Andalusia
  - Consulta privada Dr. Rafael Cáliz, Granada, Andalusia
  - Hospital San Cecilio, Granada, Andalusia
  - Hospital Virgen de las Nieves, Granada, Andalusia
  - Hospital Quirón Málaga, Málaga, Andalusia
  - Clinica Xanit, Málaga, Andalusia
  - Consulta Dra. Belmonte, Málaga, Andalusia
  - Hospital Carlos Haya, Málaga, Andalusia
  - Hospital Virgen Macarena, Seville, Andalusia
  - Hospital Virgen del Rocío, Seville, Andalusia
  - Hospital Comarcal de Melilla, Melilla, Melilla

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Whom Fulfilled the ACR: Patients whom fulfilled the ACR 2010 criteria from 2008 to 2012, and initiated on at least one DMARD during this period.
Period: Overall Study
Arm/Group | Patients Whom Fulfilled the ACR
Started | 301
Completed | 301
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Present Adverse Events, Intolerance or Lack of Efficacy to Synthetic DMARDs That Causes a Change in Treatment Prescription When Used in Routine Clinical Practice
Time Frame: 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
percentage of participants | 65.1 [63.3 to 74.3]

2. Secondary Outcome: Percentage of Patients Who Present Adverse Events While on Treatment With Synthetic Disease-modifying Antirheumatic Drug (DMARDs) and Require a Dose Reduction of the Synthetic DMARD in Question
Time Frame: 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Patients Whom Fulfilled the ACR: Patients whom fulfilled the classification of rheumatoid arthritis (ACR) 2010 criteria from 2008 to 2012, and initiated on at least one disease-modifying antirheumatic drug (DMARD) during this period.
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
percentage of participants | 10.5 [7 to 14.9]

3. Secondary Outcome: Percentage of Patients Who Experience Adverse Events While on Treatment With Synthetic DMARDs Which Forces Drug Withdrawal
Time Frame: 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
percentage of participants | 16.1 [11.9 to 21.1]

4. Secondary Outcome: Percentage of Patients Who Require an Alternative DMARD Due to Lack of Efficacy, Defined as Primary or Secondary Failure According to the Rheumatologist In-charge of Treatment
Time Frame: 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
percentage of participants | 6.9 [4.1 to 10.7]

5. Secondary Outcome: Percentage of Patients Who Receive Subcutaneous Methotrexate
Time Frame: 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
percentage of participants | 21.2 [16.3 to 26.7]

6. Secondary Outcome: Exposure Time of Methotrexate
Description: methotrexate
Time Frame: 6 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Patients Whom Fulfilled the ACR
Number analyzed (Participants) | 301
months | 19.2 (16.5)

ADVERSE EVENTS:
Arm/Group | Patients Whom Fulfilled the ACR
Serious Adverse Events (participants affected / at risk) | 0/301
Other Adverse Events (participants affected / at risk) | 0/301

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No